CLINICAL TRIAL: NCT06722573
Title: Mechanism of Rumination in the Alleviation of Emotional Distress by Mindfulness-Based Interventions: Evidence from Behavioral Experiments
Brief Title: Mechanisms of Mindfulness Intervention：Rumination Behavioral Experiments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E20241201
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Emotional Distress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIED group (Experimental): Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge, and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression, and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version
- waitlist control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version — Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: MIED group

SUMMARY:
This study hopes to explore whether the changes in rumination exhibited in behavioral experiments mediates the effects of mindfulness intervention on alleviating emotional distress

DETAILED DESCRIPTION:
In recent years, mindfulness-based interventions (MBIs) have seen extensive application in both clinical and non-clinical settings. Studies show that mindfulness training improves emotional regulation and processing, contributing to better emotional health. MBIs have proven effective in reducing anxiety and depression among patients with conditions like multiple sclerosis, enhancing personal well-being, and alleviating chronic pain. Given the mounting evidence supporting its benefits, MBIs have become widely adopted across various settings. Nonetheless, the precise mechanisms through which mindfulness alleviates emotional distress remain poorly understood.

Rumination, a transdiagnostic process, plays a critical role in the development and persistence of emotional distress. Empirical evidence supports the effectiveness of MBIs in reducing rumination. However, the role of rumination in mediating the effects of MBIs on emotional distress remains inconsistent across studies. Kazdin (2007, 2009) outlined criteria for evaluating mechanisms and mediators, yet existing studies lack sufficient evidence to meet these standards. This study aims to explore the mechanistic role of rumination using behavioral experiments, focusing on the consistency criterion

ELIGIBILITY:
Inclusion Criteria:

* - Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.
* - Aged 18-55 years old.

Exclusion Criteria:

* - Subjects who could not access the Internet;
* - Subjects with insufficient Chinese ability;
* - Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* - Subjects with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* - Subjects with high risk of suicide.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Changes of Rumination-Reflection Questionnaire during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  Rumination-Reflection Questionnaire is a self-reported questionnaire measuring Rumination level.Scores range from 12 to 60, with higher scores indicating higher levels of Rumination.
Changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Changes of the Brief State Rumination Inventory during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  The Brief State Rumination Inventory comprises eight items designed to measure an individual's state rumination tendency at a given moment, encompassing aspects such as the intensity of negative emotions, repetitive thinking, loss of thought control, and the strength of negative affect. The total score, which is derived by summing up the scores of all items, indicates the overall level of the measured construct.
Changes of the momentary repetitive negative thinking during the intervention | pre-intervention; week 3; week 5; immediately after the intervention
  momentary repetitive negative thinking measures the "process" characteristics of rumination, which are traits that exist across diagnostic categories. The scale consists of four items (e.g., "Thoughts come to my mind that I would rather not have"). Each item focuses on a core feature of rumination - repetitiveness, intrusiveness, uncontrollability, and disruptiveness. Items are rated on a 7-point Likert scale, where 1 = not at all and 7 = extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University

IPD SHARING:
Plan to Share IPD: No